CLINICAL TRIAL: NCT02331784
Title: Plasticity-based Adaptive Cognitive Remediation for Alzheimer Disease
Acronym: PACR-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PSC-PACR-AD-01
Record Dates: First submitted 2014-12-18; First posted 2015-01-06 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Older Adults, Aging Brain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computerized Plasticity-based Software (Experimental): Computerized Plasticity-based software training requiring a total maximum of 50 treatment sessions, 4-5 times weekly, 40 minutes each session.
  Interventions: Behavioral: Computerized Plasticity-based Software
- Commercially available video game (Active Comparator): Commercially available video game training. Treatment is software based, will occur up to 50 times throughout study duration, 4-5 times per week, 40 minutes each session..
  Interventions: Behavioral: Commercially available Video Game

INTERVENTIONS:
Behavioral: Computerized Plasticity-based Software — Participants will be asked to use their assigned training program for forty minutes per session, up to five sessions per week, over 10 weeks (50 total sessions).
  Arms: Computerized Plasticity-based Software
Behavioral: Commercially available Video Game — Participants will be asked to use their assigned video games for forty minutes per session, up to five sessions per week, over 10 weeks (50 total sessions).
  Arms: Commercially available video game

SUMMARY:
The primary objective of this study is to evaluate the effects of the experimental treatment (cognitive training) further outlined in this protocol on the cognitive abilities (e.g., processing speed, attention, working memory, and executive function), brain functionality, functional status and quality of life of individuals with age-related cognitive decline as compared to a computer-based active control.

DETAILED DESCRIPTION:
The normal aging has a devastating effect on our cognitive ability to learn and remember, on the speed with which the investigators process information, and on our ability to reason. By 2050, nearly 14 million individuals in the US will be living with Alzheimer's disease (AD), up from 5 million in 2013. AD is the most common cause of dementia, resulting in the loss of cognitive functions such as memory, reasoning, language, and cognitive, social, physical, and emotional control, to the extent that losses interfere with activities of daily living and necessitate continuous monitoring and care. Many studies now show that the processing machinery of the brain is plastic and remodeled throughout life by learning and experience, enabling the strengthening of cognitive skills or abilities. Research has shown that brief, daily computerized cognitive training that is sufficiently challenging, goal-directed and adaptive enables intact brain structures to restore balance in attention and compensate for disruptions in cognitive functioning. The study aims to understand how our computer program can affect cognition and attention in those with aging brain.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65-79 years at the time of consent
2. Fluent English speakers, to ensure reasonable results neuropsychological assessments
3. Adequate sensorimotor capacity to perform the program, including visual capacity adequate to read from a computer screen at a normal viewing distance, auditory capacity adequate to understand normal speech, and motor capacity adequate to control a computer mouse
4. No evidence of dementia as indicated by Montreal Cognitive Assessment (MoCA) scores >25

Exclusion Criteria:

1. Diagnosis with Alzheimer's disease or related dementias
2. Requiring caregiver assistance in dressing/personal hygiene
3. Medical conditions predisposing to imminent functional decline
4. Recent participation of computer-delivered cognitive training
5. Diagnosis of an illness or condition with known cognitive consequences (e.g., schizophrenia, bipolar disorder, cancer, multiple sclerosis) will be excluded due to the confound with cognitive impairment from normal aging.
6. Uncorrectable acuity greater than 20/40
7. Self-reported cardiovascular disease
8. Claustrophobia or any other contraindication to MRI scanning
9. Inability to complete a 1-hour MRI
10. Any implanted devices above the waist (e.g., cardiac pacemaker or auto-defibrillators, neural pacemaker, aneurysm clips, cochlear implant, metallic bodies in the eye or central nervous system, any form of wires or metal devices that may concentrate radio frequency fields)
11. History of brain surgery; removal of brain tissue; or history of stroke.

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-04; Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Changes in performance on global cognitive composite score | Baseline and at the completion of 10 weeks of training
  Change in performance on global cognitive composite score based on the average of all normalized assessment measures.

SECONDARY OUTCOMES:
Changes in brain function | Baseline and at the completion of 10 weeks of training
  Change in resting state functional connectivity will be measured by resting State T2*weighted EPI-BOLD, a 10-minute task-free BOLD contrast sequence consisting of 300 volumes (TR=2000 ms/TE=30ms) at 3.4mm3 in-plane resolution and 3mm slice thickness. Participants will be instructed to keep their eyes open and maintain attention on a central gray fixation cross on a black screen.
Changes in brain structure | Baseline and at the completion of 10 weeks of training
  3D T1-Weighted multi-echo MPRAGE. Morphometric analyses will be based on this MRI sequence (not accelerated because the reliability of acceleration for multi-site studies has not yet been established). We will achieve spatial resolution of 1 x 1 x 1 mm voxels.
Changes in task-related brain activation | Baseline and at the completion of 10 weeks of training
  Change in functional connectivity and brain activation will be measured while performing Flanker Task.
Changes in performance on memory composite score | Baseline and at the completion of 10 weeks of training
  Change in performance on memory will be measured using the composite score created by averaging the z-scores of Visual Short Term Memory, Spatial Working Memory and N-Back tasks.
Changes in performance on executive function composite score | Baseline and at the completion of 10 weeks of training
  Change in performance on executive function will be measured using the composite score created by averaging the z-scores for the Flanker, Stroop and Trail Making tasks.
Changes in performance on processing speed composite score | Baseline and at the completion of 10 weeks of training
  Change in performance on processing speed will be measured using the composite score created by averaging the z-scores of Pattern Comparison, Letter Comparison, and Digit Symbol Coding tasks.

OTHER OUTCOMES:
Changes in Life Satisfaction | Baseline and at the completion of 10 weeks of training
  Change in life satisfaction will be measured using the age-adjusted score on General Life Satisfaction Survey from NIH Tool Box.
Changes in Perceived Stress | Baseline and at the completion of 10 weeks of training
  Change in stress will be measured using the age-adjusted score on Perceived Stress Survey from NIH Tool Box.
Changes in Self-Efficacy | Baseline and at the completion of 10 weeks of training
  Change in self-efficacy will be measured using the age-adjusted score on Self-Efficacy Survey from NIH Tool Box.
Changes in Olfaction | Baseline and at the completion of 10 weeks of training
  Changes in olfaction will be measured using the age-adjusted score on Odor Identification Test from NIH Tool Box.
Changes in Standing Balance | Baseline and at the completion of 10 weeks of training
  Changes in standing balance will be measured using age-adjusted score on Standing Balance Test from NIH Tool Box.
Change in Physical Activity | Over 10 weeks
  Change in total score based on weekly self-report dairy about physical activity over a 10 week period.
Change in Diet | Over 10 weeks
  Change in total score based on weekly self-report dairy about diet over a 10 week period.
Change in Social Activity | Over 10 weeks
  Change in total score based on weekly self-report dairy about social activity over a 10 week period.
Change in Functional Abilities | Over 10 weeks
  Change in total score based on weekly self-report dairy about functional abilities over a 10 week period

CONTACTS AND LOCATIONS:
Overall Officials: Hyunkyu Lee, Ph.D., Principal Investigator — Posit Science
Locations (1):
- University of Iowa, Iowa City, Iowa, United States